CLINICAL TRIAL: NCT05617924
Title: Comparison of the Efficacy of Conventional Physiotherapy, Mechanical Traction and Spinal Decompression Treatments in Patients With Low Back Pain
Brief Title: Efficacy of Mechanical Traction and Spinal Decompression Treatments in Patients With Low Back Pain
Status: Completed | Type: Observational
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Sevda Adar, assistant professor, Afyonkarahisar Health Sciences University
Other Study IDs: SALBP
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Low Back Pain; Lumbar Disc Disease; Lumbar Disc Herniation; Lumbar Radiculopathy; Physical Therapy
MeSH Terms: conditions — Low Back Pain; Intervertebral disc disease; Intervertebral Disc Displacement; Radiculopathy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Conventional Physiotherapy: Treatment method using physical agents such as analgesic currents and superficial-deep heaters
  Interventions: Procedure: Physical Therapy
- Mechanical Traction: It is a stretching process for the spine with a weight and pulling system for the spine.
  Interventions: Procedure: Physical Therapy
- Nonsurgical Spinal Decompression: Non-surgical spinal decompression is a technique that uses a precision computerized mechanism and opens spinal nerve roots through segmental distraction.
  Interventions: Procedure: Physical Therapy

INTERVENTIONS:
Procedure: Physical Therapy — Therapy methods using physical agents in treatment

SUMMARY:
Motorized traction and non-surgical spinal decompression treatments are relatively new treatments for which there is insufficient evidence in the literature. In this study investigators aimed to retrospectively compare the effectiveness of these treatments, which are in the field of their routine practice in their clinic.

DETAILED DESCRIPTION:
Low back pain is one of the leading causes of disability worldwide. People with physically demanding jobs, physical and mental comorbidities, smokers, and obese individuals are at greater risk for low back pain. Anatomical structures that potentially nociceptive contributors to low back pain are intervertebral discs, facet joints, and vertebral end plates. It has been determined that nonsurgical treatments are clinically effective in reducing pain and functional improvement in patients with lumbar disc herniation. However, the level of evidence has generally not been highly evaluated, which can be attributed to the paucity of well designed randomized controlled trials. Despite moderate evidence, exercise and traction are recommended. In this study investigators aimed to retrospectively compare the effectiveness of these treatments, which are in the field of their routine practice in their clinic.

01.01.2019-10.11.2022. Investigators planned to examine the records of patients aged 20-75 years who underwent physical therapy with the diagnosis of lumbar discopathy in AFSU FTR Department Physical Therapy Unit. Investigators planned to examine the routine anamnesis examination, treatment card and control evaluation records of the patients made in the FTR outpatient clinic from the automation system of their hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with lumbar disc disorders
* Patients diagnosed with lumbar vertical hernia
* Aged 20-75 years

Exclusion Criteria:

* Patients treated for acute low back pain
* Patients with a history of lumbar surgery
* Patients with Spondylolisthesis or Spinal Stenosis
* Those with inflammatory rheumatic diseases (Ankylosing spondylitis, spondylarthropathy etc.)
* Patients with sequestered hernia
* Patients with insufficient data in the records

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 20-75 who underwent physical therapy with the diagnosis of Lumbar discopathy in Afyonkarahisar Health Sciences University, Department of Physical Medicine and Rehabilitation Physical Therapy Unit between 01.01.2019-10.11.2022.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Visual Pain Scale (VAS) | 5 minutes
  Visual Pain Scale (VAS), which is easy to understand, apply and interpret, provides valid and reliable data in a short time, is the most used method in clinics. With a visual linear scale of 100 mm, the patient is told that there is no pain at the 0 point, and the most severe pain ever felt in life at the 100 point, and the patient is asked to put a mark on the point corresponding to his or her pain.
Oswestry Disability Index | 20 minutes
  The Oswestry Disability Index was first described in 1980. The questionnaire consists of 10 items addressing different aspects of the function. Each item was scored from 0 to 5, with higher values representing greater disability. The total score is multiplied by 2 and expressed as a percentage. Turkish validity and reliability have been demonstrated.

CONTACTS AND LOCATIONS:
Overall Officials: SEVDA ADAR, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Sevda Adar, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided